CLINICAL TRIAL: NCT01982526
Title: Role of Anti Mullerian Hormone for Ovarian Reserve Determination of Preoperative and Postoperative Endometrioma Patients
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ergul Demircivi Bor, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2011-84
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Endometrioma; Surgery
Keywords: Ovarian reserve; Antimullerian hormone
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — We are collecting serum samples of pre and post operative endometroma patients and measuring anti müllerian hormone levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endmetrioma surgery

SUMMARY:
Ovarian reserve influenced by many factor but especially cysts like endometrioma. Anti mullerian hormone is recent marker for ovarian reserve. The investigators are searching ovarian reserve pre and post operatively by using antimullerian hormone of endometrioma patient who are operated for their cysts.

DETAILED DESCRIPTION:
long term results of the postoperative follow up for the endometrioma patients

ELIGIBILITY:
Inclusion Criteria:

* Ultrasonographical symptomatic and benign cysts which has surgery indication.

Exclusion Criteria:

* Over 42 years old, systemic endocrine disorder, history of ovarian surgery

Ages: 17 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females who are administring gynecology clinic suffering from symptomatic benign ovarian cysts.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Long term postoperative ovarian reserve outcomes of endometrioma patients by examining antimullerian hormone. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No